CLINICAL TRIAL: NCT01831583
Title: Assessment of a New Photoplethysmographic (PPG) Method and a Pulse Arrival Time Method to Detect Upper Airway Obstruction in Patients With Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) in a Sleep Laboratory
Brief Title: Assessment of PPG & PAT to Detect Upper Airway Obstruction in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sotera Wireless, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-01
Record Dates: First submitted 2013-03-25; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Measurement of PPG waveforms (Experimental): Collection of photoplethysmograph(PPG)waveform data from patients with obstructive sleep apnea for 4-8 hours
  Interventions: Device: Measurement of PPG waveforms
- Measurement of Pulse Arrival Time (PAT) (Experimental): Collection of PAT waveform data from patients with obstructive sleep apnea for 4-8 hours
  Interventions: Device: Measurement of Pulse Arrival Time (PAT)

INTERVENTIONS:
Device: Measurement of PPG waveforms — The ViSi Vital Signs Monitor will measure PPG waveforms for 4 hours.
  Other Names: ViSi Monitor
  Arms: Measurement of PPG waveforms
Device: Measurement of Pulse Arrival Time (PAT) — The ViSi Vital Signs Monitor will measure PAT waveforms for 4 hours.
  Other Names: ViSi Monitor
  Arms: Measurement of Pulse Arrival Time (PAT)

SUMMARY:
The goal of this study is to collect raw waveform data for two separate noninvasive methods, both of which may be useful for the assessment of upper airway obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients twenty-one years of age or older

Exclusion Criteria:

* Patient refusal to participate in study
* Patients under 21 (twenty-one) years of age,
* Referring physician's refusal to have his/her patient participate in the study.
* Patients with cardiac dysrhythmia (arrhythmia), including atrial fibrillation, and frequent premature atrial and/or ventricular contractions.
* Inability to obtain a Sotera cuff pressure and/or PPG signals

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Measurement of pulse arrival time in patients with obstructive sleep apnea syndrome. | 4 - 8 hours
  The goal of this study is to collect pulse arrival time data as a means for the assessment of upper airway obstruction.

SECONDARY OUTCOMES:
Non-invasive Photoplethysmographic (PPG) measurement in patients with obstructive sleep apnea syndrome. | 4 - 8 hours
  The goal of this study is to collect PPG waveforms as a means for the assessment of upper airway obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: James Welch, MS, Study Director — Sotera Wireless
Locations (1):
- Palomar Hospital, Escondido, California, United States